CLINICAL TRIAL: NCT04560335
Title: CoachToFit: Adapted Weight Loss Intervention for Individuals With Serious Mental Illness
Brief Title: Coach to Fit Weight Loss Intervention for Individuals With Serious Mental Illness
Acronym: C2F
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 19-153
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Serious Mental Illness
Keywords: weight loss; mental illness; exercise
MeSH Terms: conditions — Weight Loss; Mental Disorders; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Methodology: The study design includes a randomized controlled trial to test the efficacy of CoachToFit and assess the hypothesized mechanisms of action. This will include enrollment of obese Veterans with SMI from the mental health clinics at one VA medical center (n=256). Individuals will be randomized to CoachToFit or usual care. Those in CoachToFit will have access to the app and coaching for 6 months. Outcomes are assessed at 6- and 12-months. Efficacy outcomes utilize objective measures. The design also includes a multi- stakeholder qualitative post-intervention evaluation guided by the RE-AIM framework to characterize factors that will inform future implementation and maintenance of CoachToFit. This will include interviews with Veterans randomized to CoachToFit (n=30); interviews with staff stakeholders (n=18); a discussion with Veterans in local Veteran groups (n=2 groups; n=11 Veterans), and interviews with national leadership (n=3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coach to fit (Experimental): CoachToFit: Those randomized to CoachToFit will have the CoachToFit app downloaded to their phone by the peer coach and will work with the coach to initialize the app. Individuals will receive an activity tracker compatible with Android OS and iOS (Amazfit Bit) and a Bluetooth scale (Smart Body scale). Participants will be instructed by the peer to complete at least two CoachToFit modules per week. Modules take about 15 minutes to complete and have embedded knowledge quizzes and end with a choice of three goals to practice over the next week. They will also set up a time for the first 20-minute coaching call, which will then continue weekly.
  Interventions: Behavioral: Coach to FIt
- Treatment as usual (Other): Veterans randomized to the treatment as usual arm will continue to access all services of the VA Pittsburgh, and will participate in three research interviews. After the first meeting, all participants will meet with a peer coach (peer specialists) who will discuss with them the importance of losing weight (using a structured conversation that follows a handout which is provided to the participant). The handout was developed with input from a VA dietitian as well as Veterans and is graphically appealing, with a simple layout, and provides information on diet and activity as well as the local MOVE! schedule
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Coach to FIt — CoachToFit: Those randomized to CoachToFit will have the CoachToFit app downloaded to their phone by the peer coach and will work with the coach to initialize the app. Individuals will receive an activity tracker compatible with Android OS and iOS (Amazfit Bit) and a Bluetooth scale (Smart Body scale). Participants will be instructed by the peer to complete at least two CoachToFit modules per week. Modules take about
  15 minutes to complete and have embedded knowledge quizzes and end with a choice of three goals to practice over the next week. They will also set up a time for the first 20-minute coaching call, which will then continue weekly.
  Arms: Coach to fit
Behavioral: Treatment as Usual — Veterans randomized to the treatment as usual arm will continue to access all services of the VA Pittsburgh, and will participate in three research interviews. After the first meeting, all participants will meet with a peer coach (peer specialists) who will discuss with them the importance of losing weight (using a structured conversation that follows a handout which is provided to the participant). The handout was developed with input from a VA dietitian as well as Veterans and is graphically appealing, with a simple layout, and provides information on diet and activity as well as the local MOVE! schedule
  Arms: Treatment as usual

SUMMARY:
This project addresses obesity in the population with SMI by evaluating a weight management program that is not only evidence-based, it is sustainable, transportable, appealing to patients, easy to use, and minimally burdensome to the healthcare system. This effort addresses two HSR&D priority areas: 1) Mental Health: Testing new models of care to improve access, cost, and/or outcomes, and 2) Health Care Informatics: Building the evidence base for ehealth/mhealth tools.

Innovation: CoachToFit's use of mobile technology is an important innovation in VA service delivery and its user-centered design involving individuals with SMI was the first of its kind. CoachToFit is enhanced by data visualization in real-time via a web-based dashboard used by VA peer specialists and their supervisor. The Investigators are aware of no other evidence-based mobile platforms to help people with SMI reduce their weight

DETAILED DESCRIPTION:
Between 40% to 60% of individuals with serious mental illness (SMI) are obese. Obesity and physical inactivity result in increased rates of chronic diseases, increased risk of death, and substantial health care costs. Treatment guidelines recommend that individuals with SMI who are overweight should be offered evidence-based weight loss interventions, including psychosocial interventions. The VA's weight management program, MOVE!, is attended by less than 5% of the overweight population and is not adapted to the cognitive needs and patient preferences for the population with SMI. Effective adapted weight management programs are not offered in VA because the programs are time-intensive and require the skills of trained providers who are often in short-supply. CoachToFit can address this gap in care. CoachToFit is a weight management program, adapted for the population with SMI, that includes a smartphone app delivering evidence-based weight management services with weekly telephonic support from a VA peer specialist who acts as a wellness coach. Peer specialists are individuals who draw upon lived experiences with SMI to provide services to others with SMI in clinical settings. CoachToFit was shown to have high rates of acceptability and usability and was efficacious for weight loss in a small sample. VA has an opportunity to address obesity in the population with serious mental illness, currently a substantial gap in care.

Significance/Impact: This project addresses obesity in the population with SMI by evaluating a weight management program that is not only evidence-based, it is sustainable, transportable, appealing to patients, easy to use, and minimally burdensome to the healthcare system. This effort addresses two HSR&D priority areas: 1) Mental Health: Testing new models of care to improve access, cost, and/or outcomes, and 2) Health Care Informatics: Building the evidence base for ehealth/mhealth tools.

Innovation: CoachToFit's use of mobile technology is an important innovation in VA service delivery and its user-centered design involving individuals with SMI was the first of its kind. CoachToFit is enhanced by data visualization in real-time via a web-based dashboard used by VA peer specialists and their supervisor. The investigators are aware of no other evidence-based mobile platforms to help people with SMI reduce their weight.

ELIGIBILITY:
Inclusion Criteria:

* chart diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or recurrent major depressive disorder with psychosis;
* age 18 and over;
* BMI >= 30.0 (obese); and
* ownership of a phone running Android OS or iOS (iPhone).

Exclusion Criteria:

* chart diagnosis of dementia;
* history of bariatric surgery;
* pregnant and nursing mothers;
* patient has a conservator/legally authorized representative who makes their medical decisions;
* psychiatric hospitalization during the month prior to enrollment.

Additionally, we will follow the American College of Sports Medicine recommendations for health screening and risk stratification in preparation for starting a moderate intensity exercise program to ensure that participants enrolled are capable of safely engaging in the app's recommendations regarding physical activity. Specifically, all potential participants will be given the Physical Activity Readiness Questionnaire (PAR-Q), a screening tool often used in weight management trials. If they endorse symptoms or major signs suggestive of cardiopulmonary disease (i.e., angina, anginal equivalent, dyspnea, syncope, orthopnea, edema, palpitations or claudication), which is a score >=1 on the PAR-Q, they will need clearance from a VA physician before enrolling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
EATING HABITS CONFIDENCE SURVEY | Change from Baseline to 6 months and baseline to 12 months
  Measures a participants confidence in their eating habits and potential for change. 32 items. Scale is 1 to 5. Total score ranges from 32 to 160, with higher scores meaning more confidence in changing to healthy eating habits.
Measure Usability and Acceptability | 6 month interview
  Measures attitudes towards the Coach to fit intervention. 10 items. Scale is 1 = strongly disagree to 5 = strongly agree. After some calculations, total score ranges from 1- 100, with higher scores meaning more acceptability.
MOVE!11 Questionnaire | Change from Baseline to 6 months and baseline to 12 months
  Measures attitudes toward eating habits and weight loss. 1 item on number of minutes spent in moderate physical activity per day. higher minutes means more activity.
Weight control: Stages of change | Change from Baseline to 6 months and baseline to 12 months
  Measures willingness and readiness to change eating and exercise patterns. 4 Yes/No items. The pattern of responses places an individual into one of four categories: precontemplation (lowest), contemplation, action, maintenance (highest)
Body weight. | Change from Baseline to 6 months and baseline to 12 months
  Measurement of weight(in pounds) will be obtained for all participants using a hospital quality scale. Less pounds is better.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Chinman, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chinman M, Wang T, Dodge JR, Frank DA, McCoy JL, Cohen AN. Tailored Weight Loss Programs for Adults With Serious Mental Illness: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Dec 17:e253828. doi: 10.1001/jamapsychiatry.2025.3828. Online ahead of print. PMID 41405896

DOCUMENTS (1):
  • Informed Consent Form (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT04560335/ICF_000.pdf